CLINICAL TRIAL: NCT01418807
Title: Transumbilical Versus Transvaginal Specimen Retrieval at Minilaparoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Fabio Ghezzi, Professor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mini-LPS Specimen extraction
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain; Patients Satisfaction; Intraoperative Complications; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- TRANSVAGINAL EXTRACTION (Experimental)
  Interventions: Procedure: TRANSVAGINAL SPECIMEN EXTRACTION
- TRANSUMBILICAL EXTRACTION (Active Comparator)
  Interventions: Procedure: TRANSUMBILICAL SPECIMEN EXTRACTION

INTERVENTIONS:
Procedure: TRANSVAGINAL SPECIMEN EXTRACTION — Transvaginal specimen retrieval following posterior colpotomy
  Arms: TRANSVAGINAL EXTRACTION
Procedure: TRANSUMBILICAL SPECIMEN EXTRACTION — Transumbilical specimen retrieval following enlargement of the umbilical port
  Arms: TRANSUMBILICAL EXTRACTION

SUMMARY:
We hypothesise that pain at minilaparoscopy for gynecologic disease is reduced when transvaginal rather than transumbilical specimen extraction is accomplished. This would be due to the avoidance of a 10-mm port in the umbilicus. Visual analogue scale score of post-operative pain will be obtained and patients satisfaction will be asked at the 2-month postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* Adnexal Mass
* Benign Gynecologic Condition
* Laparoscopicb Surgery

Exclusion Criteria:

* Obliteration Of The Douglas Pouch

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology Universita' Dell'Insubria, Varese, Italy